CLINICAL TRIAL: NCT00151450
Title: An 8-Week Multicenter, Randomized, Double-Blind, Placebo-Controlled, Flexible Dose Study Of Pregabalin (300-600 Mg/Day) And Venlafaxine XR (75-225 Mg/Day) For The Acute Treatment Of DSM-IV Generalized Anxiety Disorder In Outpatients
Brief Title: Comparison of Pregabalin Versus Venlafaxine XR and Placebo in the Treatment of Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081012
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2008-03

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin
Drug: Venlafaxine XR

SUMMARY:
The purpose of the study is to compare pregabalin to Venlafaxine XR and placebo in the treatment of generalized anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients with diagnosis of generalized anxiety disorder.

Exclusion Criteria:

* Any serious or uncontrolled medical condition.
* Current diagnosis of depression, dysthymia, obsessive-compulsive disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390
Dates: Start 2005-03; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy of pregabalin and Venlafaxine XR in the treatment of generalized anxiety disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- Belgium (3):
  - Pfizer Investigational Site, De Pinte
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Waregem
- Canada (5):
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Gatineau, Quebec
  - Pfizer Investigational Site, Saint-Jean-sur-Richelieu, Quebec
- France (11):
  - Pfizer Investigational Site, Angoulême
  - Pfizer Investigational Site, Arcachon
  - Pfizer Investigational Site, Bully-les-Mines
  - Pfizer Investigational Site, Cherbourg
  - Pfizer Investigational Site, Élancourt
  - Pfizer Investigational Site, Orvault
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Saint-André-de-Cubzac
  - Pfizer Investigational Site, Savigny-sur-Orge
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Versailles
- Pfizer Investigational Site, Bray, County Wicklow, Ireland
- Italy (4):
  - Pfizer Investigational Site, Vicenza, Bassano DEL Grappa
  - Pfizer Investigational Site, Città di Castello, Perugia
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Sassari
- Netherlands (6):
  - Pfizer Investigational Site, Wildervank, Provincie Groningen
  - Pfizer Investigational Site, Hoogvliet
  - Pfizer Investigational Site, Huizen
  - Pfizer Investigational Site, Losser
  - Pfizer Investigational Site, Musselkanaal
  - Pfizer Investigational Site, Oude Pekela
- Spain (8):
  - Pfizer Investigational Site, Vic, Barcelona
  - Pfizer Investigational Site, Alcalá de Henares, Madrid
  - Pfizer Investigational Site, Langreo, Principality of Asturias
  - Pfizer Investigational Site, Gandia, Valencia
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Salamanca
  - Pfizer Investigational Site, Zamora
- Sweden (7):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Sundsvall
  - Pfizer Investigational Site, Trollhättan

REFERENCES:
- [Derived] Kasper S, Herman B, Nivoli G, Van Ameringen M, Petralia A, Mandel FS, Baldinetti F, Bandelow B. Efficacy of pregabalin and venlafaxine-XR in generalized anxiety disorder: results of a double-blind, placebo-controlled 8-week trial. Int Clin Psychopharmacol. 2009 Mar;24(2):87-96. doi: 10.1097/yic.0b013e32831d7980. PMID 21456104
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081012&StudyName=Comparison+of+Pregabalin+versus+Venlafaxine+XR+and+Placebo+in+the+Treatment+of+Generalized+Anxiety+Disorder